CLINICAL TRIAL: NCT02806297
Title: A Randomized Trial of the Effect of Timing of Cholecystectomy During Initial Admission for Mild Gallstone Pancreatitis
Brief Title: Trial of the Effect of Timing of Cholecystectomy During Initial Admission for Mild Gallstone Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Lillian Kao, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-15-0719
Record Dates: First submitted 2016-06-13; First posted 2016-06-20 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Pancreatitis
Keywords: cholecystectomy
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early cholecystectomy with IOC (Experimental): The experimental arm will be laparoscopic cholecystectomy with intraoperative cholangiogram (IOC) on admission within 24 hours of presentation regardless of whether pain or tenderness are present or laboratory values are elevated.
  Interventions: Procedure: Early cholecystectomy with IOC
- Late cholecystectomy with IOC (Active Comparator): The comparator will be laparoscopic cholecystectomy with IOC once the patient has met the following criteria: (a) a score of less than 2 on the Visual Analogue Pain Scale, (b) no tenderness on physical exam, and (c) decreased lipase to either less than half of the peak value or within normal range (73-393 U/L).
  Interventions: Procedure: Late cholecystectomy with IOC

INTERVENTIONS:
Procedure: Early cholecystectomy with IOC — The intervention will be laparoscopic cholecystectomy with intraoperative cholangiogram (IOC) on admission within 24 hours of presentation regardless of whether pain or tenderness are present or laboratory values are elevated.
  Arms: Early cholecystectomy with IOC
Procedure: Late cholecystectomy with IOC — The control will be laparoscopic cholecystectomy with IOC once the patient has met the following criteria: (a) a score of less than 2 on the Visual Analogue Pain Scale, (b) no tenderness on physical exam, and (c) decreased lipase to either less than half of the peak value or within normal range (73-393 U/L).
  Arms: Late cholecystectomy with IOC

SUMMARY:
Randomized trial of laparoscopic cholecystectomy with cholangiogram on admission versus after resolution of pain for mild gallstone pancreatitis.

DETAILED DESCRIPTION:
The purpose of this study is to perform a single-center randomized trial to compare laparoscopic cholecystectomy with intraoperative cholangiogram (IOC) within 24 hours of presentation versus after clinical resolution during index admission for mild gallstone pancreatitis on clinical and patient-reported outcomes. Additionally, this study aims to determine patients' values and preferences that influence decision-making regarding treatment options for gallstone pancreatitis. Hypothesis: During index admission for mild gallstone pancreatitis, early cholecystectomy within 24 hours of presentation regardless of symptoms or laboratory values versus after clinical resolution results in a shorter 30-day total hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gallstone pancreatitis. Patients will be considered to have gallstone pancreatitis if they have:

  1. upper abdominal pain, nausea, vomiting, and epigastric tenderness
  2. absence of ethanol abuse
  3. elevated lipase level above the upper limit of normal (>370 U/L)
  4. imaging confirmation of gallstones or sludge
* Low predicted mortality using the Bedside Index of Severity in Acute Pancreatitis (BISAP) -Diagnosis of mild pancreatitis (i.e.,no evidence of organ failure or local or systemic complications)
* Scheduled for laparoscopic cholecystectomy prior to discharge
* Lack of any very strong indicator for choledocholithiasis based on the American Society for Gastrointestinal Endoscopy (ASGE) guidelines
* Clinical stability as denoted by admission to a non-monitored floor bed.

Exclusion criteria

* Pregnancy
* Severe preexisting medical comorbidities precluding surgery, organ failure, local or systemic complications of acute pancreatitis
* Chronic pancreatitis
* Native language other than English and Spanish
* Patient refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-08-11 (Actual)

PRIMARY OUTCOMES:
30-day hospital length of stay | 30 days

SECONDARY OUTCOMES:
Time from admission to cholecystectomy | up to 10 days
Initial hospital LOS | up to 30 days
Number of participants who underwent conversion to open cholecystectomy | 30 days
Change in patient reported outcomes as assessed by the Gastrointestinal Quality-of-Life Index (GIQLI) | baseline, 1 week
Change in patient reported outcomes as assessed by the Gastrointestinal Quality-of-Life Index (GIQLI) and Patients' Experience of Surgery Questionnaire (PESQ) | baseline, 6 weeks
Change in patient reported outcomes as assessed by the Patients' Experience of Surgery Questionnaire (PESQ) | baseline, 1 week
Change in patient reported outcomes as assessed by the Patients' Experience of Surgery Questionnaire (PESQ) | baseline, 6 weeks
Change in health-related quality of life as assessed by the standard gamble | baseline, 1 week
Change in health-related quality of life as assessed by the standard gamble | baseline, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lillian S Kao, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Lyndon B. Johnson General Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Mueck KM, Wei S, Pedroza C, Bernardi K, Jackson ML, Liang MK, Ko TC, Tyson JE, Kao LS. Gallstone Pancreatitis: Admission Versus Normal Cholecystectomy-a Randomized Trial (Gallstone PANC Trial). Ann Surg. 2019 Sep;270(3):519-527. doi: 10.1097/SLA.0000000000003424. PMID 31415304
- [Derived] Mueck KM, Wei S, Liang MK, Ko TC, Tyson JE, Kao LS. Protocol for a randomized trial of the effect of timing of cholecystectomy during initial admission for predicted mild gallstone pancreatitis at a safety-net hospital. Trauma Surg Acute Care Open. 2018 Jan 20;3(1):e000152. doi: 10.1136/tsaco-2017-000152. eCollection 2018. PMID 29766134